CLINICAL TRIAL: NCT07342985
Title: Impact of Medicalized Residential Care (LAM) on the Development of Care Plans for Vulnerable Patients in Palliative Care: a Qualitative Study
Brief Title: Impact of Medicalized Residential Care (LAM) on the Development of Care Plans for Vulnerable Patients in Palliative Care
Acronym: LAM-SP
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9817
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Palliative Care
Keywords: Palliative care; Palliative care pathology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the research is to identify the factors influencing the development of care plans for vulnerable patients admitted to medicalized care facilities (LAM) and in palliative care.

ELIGIBILITY:
Inclusion Criteria:

* Adult subject (≥18 years old)
* Subject residing in one of the two LAM regions of Alsace (France) at the time of the study and suffering from a palliative-care condition (the nature of the condition (or conditions) is not specified)

Exclusion Criteria:

- Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subject residing in one of the two LAM regions of Alsace and suffering from a palliative-care condition (the nature of the condition (or conditions) is not specified)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10-10 (Estimated)

PRIMARY OUTCOMES:
Analysis of Interviewees' Discourse Regarding the Organizational, Human, and Relational Resources Implemented Within the Facilities to Develop a Care Plan | Up to 12 months
  There is no evaluation in this study: it simply aims to identify the factors influencing the development of care plans for vulnerable patients requiring palliative care and admitted to medical facilities (LAM)

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Accompagnement et de Soins Palliatifs - CHU de Strasbourg - France, Strasbourg, France